CLINICAL TRIAL: NCT00343525
Title: A Phase Ib Open-Label, Escalating Repeat-Dose Trial of Bavituximab (Chimeric Anti-Phosphatidylserine Monoclonal Antibody) in Patients With Chronic Hepatitis C
Brief Title: Repeat-Dose Study of Bavituximab in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Dianne Uphoff/Senior Clinical Project Manager, Peregrine Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 0601
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-04

CONDITIONS: Hepatitis C
Keywords: HCV; monoclonal antibody; phase 1
MeSH Terms: conditions — Hepatitis C | interventions — bavituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bavituximab

SUMMARY:
The purpose of this study is to determine the safety and tolerability of bavituximab when administered via an arm vein as multiple infusions and to examine how bavituximab behaves in the body and how it effects the amount of hepatitis C virus and immune modulators in individuals with chronic infection.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a world wide public health concern and is the most common chronic bloodborne infection in the United States and the leading indication for liver transplantation. Laboratory and animal studies have demonstrated that bavituximab binds viruses and virally infected cells and prolongs survival in lethally infected animals. This study will examine the safety and tolerability of bavituximab when administered as multiple infusions to patients with chronic HCV infection. Groups of patients will be treated with escalating doses of bavituximab twice weekly for 2 weeks and followed for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Chronic Hepatitis C infection based on history and detectable serum HCV RNA including treatment naïve subjects as well as subjects who are partial responders and/or relapsers to prior therapy(ies)
* All genotypes of HCV acceptable
* Complete Blood Counts within normal limits
* Normal renal function (serum creatinine within normal limits)
* Normal coagulation profile (PT/INR and aPTT within normal limits)
* Patients of reproductive potential must agree to use an approved form of barrier contraception. Female patients must have a negative serum pregnancy test at prestudy (not applicable to patients with bilateral oophorectomy and/or hysterectomy or to those patients who are postmenopausal)

Exclusion Criteria:

* Prior exposure to any chimeric antibody
* Any other cause of liver disease other than chronic hepatitis C, such as autoimmune or alcoholic liver disease.
* Decompensated clinical liver disease, including a history of prolonged clotting times, hypoalbuminemia, encephalopathy, treatment for elevated ammonia levels, or ascites
* Any evidence of clinically significant bleeding defined as gross hematuria, hemoptysis, or gastrointestinal bleeding
* Known history of bleeding diathesis or coagulopathy (e.g., von Willebrand Disease or Hemophilia)
* Any history of thromboembolic events [e.g., deep vein thrombosis (DVT) or pulmonary thromboembolism (PE)] including central venous catheter-related thrombosis within the past 12 months
* Concurrent therapy with oral or parenteral anticoagulants
* Concurrent hormone therapy (i.e., estrogen contraceptives, hormone replacement, anti-estrogen)
* Antiviral therapy within 4 weeks of day 0
* Investigational therapy within 4 weeks of day 0
* Major surgery within 4 weeks of day 0
* Pregnant or nursing women
* Uncontrolled intercurrent disease (e.g., diabetes, hypertension, thyroid disease)
* Any history of angina pectoris, coronary artery disease or cerebrovascular accident, or transient ischemic attack
* A history of any condition requiring anti-platelet therapy with the exception of general cardiovascular prophylaxis with aspirin
* A history of any condition requiring treatment (past or current) with coumarin-type agents
* Cardiac arrhythmia requiring medical therapy
* Serious non-healing wound (including wound healing by secondary intention, ulcer, or bone fracture)
* Requirement for chronic daily treatment with NSAIDs, antiplatelet drugs (e.g., phosphodiesterase inhibitors, adenosine diphosphate receptor antagonists), or steroids
* Cancer, autoimmune disease or any disease or concurrent therapy known to cause significant alteration in immunologic function
* Known chronic infection with HIV or HBV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-05; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
adverse events
laboratory evaluations
human anti-chimeric antibody
pharmacokinetic analysis
viral kinetic analysis
cytokine analysis

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lawitz, MD, Principal Investigator — Alamo Medical Research; Eliot W Godofsky, MD, Principal Investigator — University Hepatitis Center
Locations (2):
- United States (2):
  - University Hepatitis Center at Bach & Godofsky MD PA, Sarasota, Florida
  - Alamo Medical Research, San Antonio, Texas